CLINICAL TRIAL: NCT05893069
Title: Ability of Oral Oxandrolone to Aid in Rehabilitation and Outcomes of Multiligament Knee Reconstructions: A Double-Blind, Randomized Controlled Trial
Brief Title: Oxandrolone Multiligament Knee
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: FDA withdrew approval of the study product
Sponsor: George F. Hatch (Other)
Responsible Party: Sponsor-Investigator, George F. Hatch, Associate Professor, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HS-20-00161
Record Dates: First submitted 2023-05-16; First posted 2023-06-07 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Ligament Tear Knee
Keywords: Oxandrolone; Testosterone; Anabolic Steroid
MeSH Terms: interventions — Oxandrolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Oxandrolone
  Interventions: Drug: Oxandrolone
- Placebo Group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxandrolone — oral oxandrolone for 12 weeks
  Arms: Treatment group
Drug: Placebo — oral placebo for 12 weeks
  Arms: Placebo Group

SUMMARY:
This study is about healing after a rmultiligament knee reconstruction procedure. We hope to learn if a biologic medication: Oxandrolone, a synthetic derivative of the human hormone Testosterone (the principal male sex hormone and an anabolic steroid), given for 12 weeks is effective in aiding in the healing process and restoring muscle mass.

ELIGIBILITY:
Inclusion Criteria:

• Patients with MRI proven multiligament knee injury scheduled to undergo multiligament knee reconstruction

Exclusion Criteria:

* Patients with prior ipsilateral knee surgery
* Untreated diabetes mellitus
* Pituitary tumor
* Rheumatoid Arthritis
* Uncontrolled hypertension
* Congestive Heart Failure
* Myocardial Infarction within the past 6 months
* End-stage renal disease
* Liver enzymes two times the normal value
* DVT within the past 6 months
* Disorder of the coagulation system
* Currently taking anticoagulation
* Prior or current use of anabolic steroids
* Chromosomal disorders
* Prostate cancer
* Breast cancer
* Hypercalcemia
* Patients with COPD not responsive to bronchodilators
* Patients with known liver disease
* Patients at risk for liver tumors
* Severe hyperlipidemia
* Patients taking medications that interfere with testosterone production or function, including but not limited to 5α-reductase inhibitors, acetaminophen (Tylenol, others), cholesterol lowering

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
lean body mass | Change from baseline at 52 weeks
  measured by bioelectrical impedance analysis
body fat percentage | Change from baseline at 52 weeksf
  measured by bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: George Hatch, MD, Principal Investigator — University of Southern California
Locations (1):
- Keck School of Medicine of the University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No